CLINICAL TRIAL: NCT00418886
Title: A Phase III, Randomized, Double-blinded, Parallel Group, Multi-centre Study to Assess the Efficacy and Safety of ZD6474 (ZACTIMA™) in Combination With Pemetrexed (Alimta®) Versus Pemetrexed Alone in Patients With Locally-Advanced or Metastatic NSCLC
Brief Title: Efficacy Study Comparing ZD6474 in Combination With Pemetrexed and Pemetrexed Alone in 2nd Line NSCLC Patients
Acronym: ZEAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00036; EUDRACT No. 2006-003695-35; LPS15296 (Other: Sanofi)
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — vandetanib; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Placebo Vandetanib + Pemetrexed
  Interventions: Drug: Pemetrexed
- 2 (Experimental): Vandetanib + Pemetrexed
  Interventions: Drug: Vandetanib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Vandetanib — oral once daily tablet
  Other Names: ZACTIMA™; ZD6474; SAR390530
  Arms: 2
Drug: Pemetrexed — intravenous infusion
  Other Names: Pemetrexed disodium; Alimta®

SUMMARY:
Non-small cell lung cancer (NSCLC) can be treated with drugs that kill tumour cells, stop them from dividing, or stop the growth of the blood supply that cancers need to grow and spread. Clinical research has shown that drugs that inhibit vascular endothelial growth factor receptor (VEGFR) or epidermal growth factor receptor (EGFR) signalling can increase overall survival in patients with advanced non-small cell lung cancer (NSCLC). Preclinical studies have shown that vandetanib (ZD6474) is an inhibitor of both VEGFR and EGFR signalling. Giving vandetanib may therefore inhibit the growth of cancer cells by blocking their blood supply and by stopping them from dividing. This lung cancer study is to investigate if adding vandetanib to Alimta (pemetrexed) is more effective than Alimta (pemetrexed) alone.

DETAILED DESCRIPTION:
This randomized phase III non-small cell lung cancer clinical trial is studying the effect of Alimta (pemetrexed) plus vandetanib to see how well the combination works compared to Alimta (pemetrexed) alone in patients who have previously been treated for non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Female or male aged 18 years or above
* Histologic or cytologic confirmation of locally advanced or metastatic NSCLC (stage IIIB or IV) on entry into study
* Failure of 1st line anti-cancer therapy (either radiological documentation of disease progression or due to toxicity) or subsequent relapse of disease following 1st line therapy
* WHO Performance status 0 - 2
* One or more measurable lesions at least 10 mm in the longest diameter (LD) by spiral CT scan or 20 mm with conventional techniques according to RECIST criteria. Previously irradiated lesions will not be considered measurable.
* Life expectancy of 12 weeks or longer
* Negative pregnancy test for women of childbearing potential only

Exclusion Criteria:

* Mixed small cell and non-small cell lung cancer histology
* Patients have received 2nd-line or subsequent anti-cancer therapy
* Prior treatment with pemetrexed
* Prior treatment with VEGFR TKIs (previous treatment with bevacizumab [Avastin] is permitted)
* Known or suspected brain metastases or spinal cord compression, unless treated at least 4 weeks before entry, and stable without steroid treatment for 10 days
* The last radiation therapy within 4 weeks before the start of study therapy, not including local palliative radiation
* The last dose of prior chemotherapy or other anti-cancer therapy is discontinued less than 3 weeks before the start of study therapy (6 weeks for nitrosoureas, mitomycin, and suramin)
* Major surgery within 4 weeks before entry, or incompletely healed surgical incision
* Neutrophils <1.5 x 109/L or platelets <100 x 109/L
* Serum bilirubin >1.5 x the upper limit of reference range (ULRR)
* Creatinine clearance <50 ml/min calculated by either Cockcroft -Gault, 24 hours urine collection, EDTA scan or other validated methods
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULRR in the absence of liver metastases, or > 5 x ULRR in the presence of liver metastases
* Alkaline phosphatase (ALP) >2.5 x ULRR in the absence of liver metastases, or >5 x ULRR in the presence of liver metastases
* Current active gastrointestinal disease that may affect the ability of the patient to absorb ZD6474 or tolerate diarrhoea
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol
* Any unresolved toxicity greater than CTCAE Grade 2 from previous anti-cancer therapy
* Significant cardiovascular event (e.g., myocardial infarction, superior vena cava [SVC] syndrome), New York Heart Association [NYHA] classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* QT prolongation with other medications that required discontinuation of that medication
* Presence of left bundle branch block (LBBB)
* QTc with Bazett's correction unmeasurable or ≥ 480 msec on screening ECG (Note: If a patient has QTc interval ≥480 msec on screening ECG, the screen ECG may be repeated twice [at least 24 hours apart]. The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study) Patients who are receiving a drug that has a risk of QTc prolongation are eligible if QTc is <460 msec.
* Potassium <4.0 mmol/L despite supplementation; serum calcium (or ionized or adjusted for albumin), or magnesium out of normal range despite supplementation
* Women who are pregnant or breast-feeding
* Any concomitant medications that may cause QTc prolongation or induce Torsades de Pointes or induce CYP3A4 function. Drugs that have a risk of QTc prolongation, that in the investigator's opinion cannot be discontinued, are allowed, but only of the QTc is <460 msec
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 millimetre of mercury [mmHg] or diastolic blood pressure greater than 100 mmHg)
* Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix and adequately treated basal cell or squamous cell carcinoma of the skin
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment
* Concomitant use of yellow fever vaccine or any live attenuated vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (110):
- United States (23):
  - Research Site, Casa Grande, Arizona
  - Research Site, Chandler, Arizona
  - Research Site, Farmington, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Orlando, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Skokie, Illinois
  - Research Site, Sioux City, Iowa
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Mineola, New York
  - Research Site, Rochester, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Salt Lake City, Utah
- Argentina (8):
  - Research Site, Avellaneda
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Ramos Mejía
  - Research Site, Salta
  - Research Site, Santa Fe
- Australia (7):
  - Research Site, Chermside
  - Research Site, Fitzroy
  - Research Site, Footscray
  - Research Site, Heidelberg
  - Research Site, Randwick
  - Research Site, St Leonards
  - Research Site, Wodonga
- Belgium (3):
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Leuven
  - Research Site, Liège
- Colombia (4):
  - Research Site, Bogotá
  - Research Site, Medellín
  - Research Site, Pereira
  - Research Site, Valledupar
- France (5):
  - Research Site, Avignon
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Pontoise
  - Research Site, Strasbourg
- Germany (5):
  - Research Site, Cologne
  - Research Site, Hanover
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Leipzig
- Greece (3):
  - Research Site, N. Faliro
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- India (2):
  - Research Site, Ahmedabad
  - Research Site, Vellore
- Israel (8):
  - Research Site, Beer-Sheeva
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Safed
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (5):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Roma
  - Research Site, S.Andrea Delle Fratte
- Mexico (3):
  - Research Site, Aguascalientes
  - Research Site, México
  - Research Site, Puebla City
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Pasay
  - Research Site, Quezon City
- Portugal (3):
  - Research Site, Lisbon
  - Research Site, Santa Maria da Feira
  - Research Site, Setúbal
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Lugo
  - Research Site, Majadahonda
  - Research Site, Mataró(Barcelona)
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Santiago de Compostela(A Coru
  - Research Site, Vigo(Pontevedra)
- Sweden (5):
  - Research Site, Lund
  - Research Site, Sundsvall
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Västerås
- Research Site, Taipei, Taiwan
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, Leeds
  - Research Site, Manchester
  - Research Site, Wolverhampton
- Venezuela (2):
  - Research Site, Caracas
  - Research Site, Valencia

REFERENCES:
- [Result] de Boer RH, Arrieta O, Yang CH, Gottfried M, Chan V, Raats J, de Marinis F, Abratt RP, Wolf J, Blackhall FH, Langmuir P, Milenkova T, Read J, Vansteenkiste JF. Vandetanib plus pemetrexed for the second-line treatment of advanced non-small-cell lung cancer: a randomized, double-blind phase III trial. J Clin Oncol. 2011 Mar 10;29(8):1067-74. doi: 10.1200/JCO.2010.29.5717. Epub 2011 Jan 31. PMID 21282537
- [Derived] Platt A, Morten J, Ji Q, Elvin P, Womack C, Su X, Donald E, Gray N, Read J, Bigley G, Blockley L, Cresswell C, Dale A, Davies A, Zhang T, Fan S, Fu H, Gladwin A, Harrod G, Stevens J, Williams V, Ye Q, Zheng L, de Boer R, Herbst RS, Lee JS, Vasselli J. A retrospective analysis of RET translocation, gene copy number gain and expression in NSCLC patients treated with vandetanib in four randomized Phase III studies. BMC Cancer. 2015 Mar 23;15:171. doi: 10.1186/s12885-015-1146-8. PMID 25881079
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=341&filename=CSR-D4200C00036.pdf
- See also: CSR-D4200C00036.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=341&filename=CSR-D4200C00036.pdf
- See also: Vandetanib_study_36_ZEAL_CSP_redacted_SECURE — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=341&filename=Vandetanib_study_36_ZEAL_CSP_redacted_SECURE.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled 09 January 2007, last participant enrolled 29 February 2008, cut off date 05 September 2008.
Pre-assignment Details: A total of 534 participants were randomized in the study.
Groups:
- Vandetanib Plus Pemetrexed: Vandetanib [100 milligram (mg) daily] plus pemetrexed [500 mg/meter square (m^2) given on Day 1 of each 21-day cycle].
- Placebo Plus Pemetrexed: Placebo plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle).
Period: Randomized Period
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Started | 256 (Randomized participants.) | 278 (Randomized participants.)
Treated | 260 (Four participants randomized to the "Placebo Plus Pemetrexed" reporting group were erroneously assigned to receive vandetanib during the Randomized Period.) | 273
Completed | 30 (Ongoing study treatment at data cut-off.) | 23 (Ongoing study treatment at data cut-off.)
Not Completed | 226 | 255
Not completed — discontinue treatment survival follow-up | 90 | 91
Not completed — Death | 122 | 147
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Lost to Follow-up | 4 | 6
Not completed — withdrawn due to other reason | 1 | 0
Not completed — randomised but no treatment received | 0 | 1
Period: Survival Follow-up Period
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Started | 120 (Completed randomization treatment, discontinue treatment survival follow-up, and took vandetanib from placebo group.) | 114 (Completed randomization treatment, discontinue treatment survival follow-up, and minus 4 who took vandetanib.)
Treated With Vandetanib | 124 (Four participants randomized to the "Placebo Plus Pemetrexed" reporting group were erroneously assigned to receive vandetanib during the Randomized Period.) | 110
Completed (Participants with end of treatment or death due to any cause.) | 120 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Vandetanib Plus Pemetrexed: Vandetanib (100 mg daily) plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle).
- Total: Total of all reporting groups
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed | Total
Number analyzed (Participants) | 256 | 278 | 534
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (9.95) | 60.2 (9.5) | 59.4 (9.73)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 97 | 107 | 204
  Male | 159 | 171 | 330

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in the Overall Population
Description: Median time (in weeks) from randomization until objective disease progression or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable Response Evaluation Criteria in Solid Tumors (RECIST) assessment.
Time Frame: RECIST tumour assessments carried out every 6 weeks (+/- 3 days) from randomization until objective progression
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
weeks | 17.6 [13.4 to 18.9] | 11.9 [11.4 to 15.9]

2. Primary Outcome: Progression-Free Survival in the Female Population
Description: Median time (in weeks) from randomization until objective disease progression or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment.
Time Frame: RECIST tumour assessments carried out every 6 weeks (+/- 3 days) from randomization until objective progression
Population: The female analysis set included all randomized female participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 97 | 107
weeks | 17.9 [14.7 to 22.7] | 13.0 [11.1 to 17.7]

3. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from date of randomization until death. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive (i.e, their status must be known at the censored date and should not be lost to follow up or unknown).
Time Frame: Time to death in months
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
months | 10.5 [8.9 to 12.3] | 9.2 [7.1 to 12.0]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of participants that are responders i.e, those participants with a confirmed best objective response of complete response (CR) or partial response (PR) as defined by RECIST criteria. The categories for best objective response are CR, PR, stable disease (SD)>= 6 weeks, progressive disease (PD) or NE.
Time Frame: Each participant was assessed for objective response from the sequence of RECIST scan data up to data cut off. RECIST tumour assessments carried out every 6 weeks (+/- 3 days) from randomization until objective progression
Population: The full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
percentage of participants | 19.1 | 7.9

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR is defined as the number of patients who achieved disease control at 6 weeks following randomization. Disease control at 6 weeks is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 6 weeks.
Time Frame: RECIST tumour assessments carried out every 6 weeks (+/- 3 days) from randomization until objective progression
Population: The full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
percentage of participants | 56.6 | 45.7

6. Secondary Outcome: Duration of Response (DoR)
Description: Response is defined as a confirmed best objective response of CR or PR. Duration of response is defined as time from the date of first documented response until date of documented progression or death in the absence of disease progression (provided death is within 3 months of last RECIST assessment).
Time Frame: RECIST tumour assessments carried out every 6 weeks (+/- 3 days) from randomization until objective progression
Population: The full analysis set included all randomized participants. Only participants with response are analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 49 | 22
weeks | 24.1 [17.4 to 30.0] | 24.4 [18.0 to 32.0]

7. Secondary Outcome: Time to Deterioration of Disease-Related Symptoms (TDS) by Lung Cancer Symptom Scale (LCSS) Total Score
Description: TDS is the interval from the date of randomization to the first assessment of worsened without an improvement in the next 21 days. A deterioration in symptoms is defined as a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 21 days. The LCSS scale measures changes in symptoms associated with lung cancer.
Time Frame: LCSS questionnaires are to be administered every 3 weeks after randomization
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
weeks | 18.1 [15.1 to 23.6] | 12.1 [9.7 to 17.3]

8. Secondary Outcome: Time to Deterioration of Disease-Related Symptoms by Average Symptom Burden Index (ASBI) Score
Description: Time to deterioration is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 21 days. A deterioration in symptoms is defined as a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 21 days. The ASBI is derived from 6 of LCSS's 9 items.
Time Frame: ASBI is a score taken from the LCSS questionnaires which are to be administered every 3 weeks after randomization
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
weeks | 16.0 [14.0 to 20.3] | 13.4 [10.3 to 17.9]

9. Secondary Outcome: Longitudinal Analysis of Lung Cancer Symptom Scale Total Score
Description: The longitudinal data analysis will include all non-missing visit scores and the model will include only the first 12 weeks of data. LCSS total score is an average of all 9 visual analogue participant scales from "none" [0 millimeter (mm)] to "as much as it could be" (100 mm).
Time Frame: LCSS questionnaires are to be administered every 3 weeks after randomization
Population: The full analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mms on a visual analogue scale
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
mms on a visual analogue scale | 25.7 (2.85) | 28.3 (2.77)

10. Secondary Outcome: Longitudinal Analysis of Average Symptom Burden Index Score
Description: The longitudinal data analysis will include all non-missing visit scores and the model will include only the first 12 weeks of data. ASBI is an average of the 6 symptom visual analogue patient scales from "none" (0 mm) to "as much as it could be" (100 mm).
Time Frame: ASBI is a score taken from the LCSS questionnaires administered every 3 weeks after randomization
Population: The full analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mms on a visual analogue scale
Arm/Group | Vandetanib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 256 | 278
mms on a visual analogue scale | 21.7 (2.75) | 24.3 (2.67)

ADVERSE EVENTS:
Time Frame: From the date of informed consent up to the study completion for each participant, approximately 193 months.
Description: The Safety analysis set included all participants who received at least 1 dose of vandetanib or placebo. Four participants randomized to the "Placebo Plus Pemetrexed" reporting group were erroneously assigned to receive vandetanib during the Randomized Period. Therefore, the total number of participants received the Vandetanib Plus pemetrexed treatment was 260 whereas the total participants received "Placebo Plus Pemetrexed" were 273 during the Randomized Period.
Groups:
- Randomized Period: Vandetanib Plus Pemetrexed: Vandetanib (100 mg daily) plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle) in randomized period.
- Randomized Period: Placebo Plus Pemetrexed: Placebo plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle) in randomized period.
- Survival Follow-up Period: Vandetanib Plus Pemetrexed: Vandetanib (100 mg daily) plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle) in survival follow-up period.
- Survival Follow-up Period: Placebo Plus Pemetrexed: Placebo plus pemetrexed (500 mg/m^2 given on Day 1 of each 21-day cycle) in survival follow-up period.
Arm/Group | Randomized Period: Vandetanib Plus Pemetrexed | Randomized Period: Placebo Plus Pemetrexed | Survival Follow-up Period: Vandetanib Plus Pemetrexed | Survival Follow-up Period: Placebo Plus Pemetrexed
All-Cause Mortality (participants affected / at risk) | 122/260 | 147/273 | 63/124 | 58/110
Serious Adverse Events (participants affected / at risk) | 84/260 | 94/273 | 7/124 | 3/110
Other Adverse Events (participants affected / at risk) | 234/260 | 242/273 | 22/124 | 19/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Period: Vandetanib Plus Pemetrexed (N=260) | Randomized Period: Placebo Plus Pemetrexed (N=273) | Survival Follow-up Period: Vandetanib Plus Pemetrexed (N=124) | Survival Follow-up Period: Placebo Plus Pemetrexed (N=110)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (8) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reflux Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (8) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organ Failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Performance Status Decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (9) | 3 (4) | 0 (0) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 10 (13) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaesthetic Complication Cardiac (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Artery Embolism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Prerenal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 10 (10) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Pulmonary Fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena Cava Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Period: Vandetanib Plus Pemetrexed (N=260) | Randomized Period: Placebo Plus Pemetrexed (N=273) | Survival Follow-up Period: Vandetanib Plus Pemetrexed (N=124) | Survival Follow-up Period: Placebo Plus Pemetrexed (N=110)
Anaemia (Blood and lymphatic system disorders) | 19 (27) | 54 (59) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 18 (27) | 17 (22) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 21 (32) | 26 (35) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 12 (12) | 14 (16) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 16 (21) | 15 (17) | 1 (1) | 2 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 14 (16) | 17 (18) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 52 (69) | 53 (65) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 66 (95) | 48 (66) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 21 (25) | 11 (11) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 73 (100) | 98 (167) | 0 (0) | 3 (12)
Stomatitis (Gastrointestinal disorders) | 19 (25) | 18 (24) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 37 (42) | 55 (97) | 3 (3) | 3 (10)
Asthenia (General disorders) | 29 (34) | 43 (63) | 4 (4) | 2 (2)
Fatigue (General disorders) | 99 (127) | 118 (159) | 2 (2) | 2 (2)
Oedema Peripheral (General disorders) | 11 (12) | 22 (24) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 25 (32) | 43 (60) | 2 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 12 (14) | 14 (19) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 23 (23) | 15 (15) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 56 (72) | 65 (82) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 16 (17) | 2 (2) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 24 (25) | 31 (32) | 1 (1) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 21 (26) | 2 (2) | 3 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 23 (25) | 1 (1) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 18 (18) | 0 (0) | 4 (4)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (18) | 21 (24) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 20 (26) | 23 (30) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 28 (35) | 40 (50) | 1 (1) | 3 (4)
Anxiety (Psychiatric disorders) | 11 (12) | 16 (16) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 14 (14) | 17 (17) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 34 (38) | 27 (27) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (75) | 59 (68) | 4 (4) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 6 (6) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 (53) | 56 (60) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 12 (15) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 17 (21) | 1 (1) | 1 (3)
Acne (Skin and subcutaneous tissue disorders) | 14 (15) | 8 (8) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 14 (14) | 8 (9) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 14 (18) | 12 (16) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (37) | 40 (47) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 99 (143) | 71 (93) | 3 (5) | 1 (1)
Hypertension (Vascular disorders) | 29 (35) | 8 (9) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.